CLINICAL TRIAL: NCT04212884
Title: Functional Decline and Quality of Life in People Aging with HIV in Asia
Brief Title: Functional Decline and QoL in People Aging with HIV in Asia
Status: Completed | Type: Observational
Sponsor: Chinese University of Hong Kong (Other)
Collaborators: University of Malaya (Other); National Taiwan University (Other); Chongqing Public Health Medical Center (Other); Tan Tock Seng Hospital (Other)
Responsible Party: Principal Investigator, Shui-Shan Lee, MD, Professor, Chinese University of Hong Kong
Other Study IDs: Geri_HIV_protocol_v4_26Nov2019
Record Dates: First submitted 2019-12-20; First posted 2019-12-30 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-02

CONDITIONS: Frailty; Disability Physical; HIV/AIDS
MeSH Terms: conditions — Frailty; Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Blood samples will be stored for future analysis of biomarkers related to inflammation and ageing.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- PLWH: PLWH followed up at the five participating HIV centers
- HIV-uninfected individuals: Age and sex-matched HIV-uninfected individuals

SUMMARY:
This is a multi-center prospective cross-sectional study to determine the burden of decline in intrinsic capacity and functional ability, and the prevalence of geriatric syndromes, such as frailty, and disability in adult people living with HIV (PLWH) in Asia.

DETAILED DESCRIPTION:
This research project is expected to have the following clinical impact

1. To understand the impact of impaired functional status in PLWH in Asia would be important to determine the long-term health burden needs in this aging population in this part of the world.
2. The identification of risk factors associated with impaired functional status would be important to guide clinical decisions in patient management, such as the choice of anti-retroviral regimen, and screening of and early intervention for modifiable risk factors. These are of paramount importance in the promotion of healthy aging in this population.
3. This proposed cross-sectional study lays the foundation for the establishment of a longitudinal cohort for long-term follow up of people aging with HIV in Asia, with the objectives of evaluating the long-term impact of aging on clinical outcomes and functional status in PLWH in this region.

ELIGIBILITY:
Inclusion Criteria:

* HIV antibody positive
* Age 35 years or above
* Asian ethnicity, including but not limited to Chinese, Malay and Indian

Exclusion Criteria:

* Inability or refusal to consent
* Active infections requiring in-hospital treatment

Min Age: 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All PLWH followed up at the five participating HIV centers will be screened and invited to participate in this study. Each site will also enroll age and sex-matched HIV-uninfected participants in a 1:2 ratio.
Sampling Method: Probability Sample
Enrollment: 1500 (Actual)
Dates: Start 2020-05-01 (Actual); Primary Completion 2025-01-31 (Actual); Study Completion 2025-01-31 (Actual)

PRIMARY OUTCOMES:
Functional disability | 24 months
  Functional disability is defined as any difficulty in any of the six areas of functioning in daily life as assessed by WHO DAS II questionnaire

SECONDARY OUTCOMES:
Composite score for intrinsic capacity | 24 months
  The score is based on (i) self-reported questions assessing the subjects' eight health domains, including mobility, self-care, cognition, interpersonal activities, vision, pain and discomfort, sleep and energy, and affect, and (ii) measures of grip strength, short physical performance battery and cognitive function
Physical performance | 24 months
  Physical performance is measured by six-metre usual gait speed. Low physical performance is defined as usual gait speed ≤0.8 m/s
Cognitive decline | 24 months
  Cognitive decline is defined as presence of HIV-associated neurocognitive disorder (HAND) according to "Frascati Criteria". Asymptomatic neurocognitive impairment (ANI) involves impairment of cognitive functioning in at least two ability domains, in the absence of interference in everyday functioning. Mild neurocognitive disorder (MND) also involves impairment in at least two ability domains, with at least mild interference in daily functioning. HIV-associated dementia (HAD) requires marked impairment in cognitive functioning in at least two ability domains, in the presence of marked impairment in day-to-day functioning
Frailty | 24 months
  Frailty is measured using the frailty index
Sarcopenia | 24 months
  Sarcopenia is defined as height-adjusted skeletal muscle mass <7.0 kg/m2 in men and 5.7 kg/m2 in women using BIA
Health-related quality of life | 24 months
  Health-related quality of life will be assessed as measured by WHO HIV BREF QOL.

CONTACTS AND LOCATIONS:
Overall Officials: Grace LUI, Principal Investigator — Chinese University of Hong Kong
Locations (2):
- Hong Kong (2):
  - Prince of Wales Hospital, Hong Kong
  - Prince of Wales Hospital, Shatin